CLINICAL TRIAL: NCT06283082
Title: Oxalate Excretion Profile in Patients with a Heterozygous Mutation of the AGXT (alanine-glyoxylate Aminotransferase) Gene - Influence of Hygienic and Dietary Conditions and Identification of Favouring Factors by Comparison of Asymptomatic and Symptomatic Patients (lithiasis or Oxalic Nephropathy)
Brief Title: Oxalate Excretion Profile in Patients with a Heterozygous Mutation of the AGXT (alanine-glyoxylate Aminotransferase) Gene
Acronym: HETEROX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_0617; ID-RCB (Other: 2023-A01406-39)
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Hyperoxaluria (Disorder)
Keywords: AGXT heterozygous mutation; lithiasis; nutrition; nephropathy
MeSH Terms: conditions — Hyperoxaluria; Lithiasis; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asymptomatic subjects with an AGXT heterozygous mutation (Experimental)
  Interventions: Diagnostic Test: Lithiasis assessment
- Symptomatic subjects with an AGXT heterozygous mutation (Active Comparator)
  Interventions: Diagnostic Test: Lithiasis assessment

INTERVENTIONS:
Diagnostic Test: Lithiasis assessment — Measurement of oxaluria and glycolaturia on 24 h urine collection, identification of lithiasis disease (biological and ultrasound) and search for lithiasis risk factors.

SUMMARY:
Primary hyperoxaluria type I (PH1) is a rare genetic disorder responsible for severe lithiasis leading to progressive deterioration of renal function and end-stage renal failure. PH1 is linked to a deficiency in glyoxylate amino transferase (AGXT), which leads to increased endogenous oxalate synthesis and hyperoxaluria. In the urine, urinary oxalate precipitates with calcium, forming insoluble crystals, leading to lithiasis and the development of nephrocalcinosis.

Non-genetic etiologies of oxalic nephropathy are well known, in particular enteric causes (malabsorptions, bypass, calcium deficiencies, etc.) and sometimes linked to increased oxalate intake in the form of nutritional or vitamin supplements, reinforcing the hypothesis of probably underestimated favouring factors of hyperoxaluria.

Until now, heterozygous patients with a mutation in the AGXT gene were considered asymptomatic. However, there have been several cases of patients with heterozygous AGXT mutations presenting with lithiasis.

Consequently, the characteristics of symptomatic and asymptomatic heterozygous patients will be studied in order to define the elements that would explain the expression of the disease (particularities of the AGXT mutation, presence of another heterozygous mutation or favorable living conditions).

The hypothesis is that there is an increase in hepatic oxalate production in heterozygous patients, which explains why they remain asymptomatic under usual conditions, but could favor stone formation under favorable conditions such as severe calcium deficiency or malabsorption.

ELIGIBILITY:
Inclusion Criteria:

* Presenting an heterozygous mutation on AGXT
* Presenting symptoms (presence or history of stones, nephrocalcinosis) or not

Exclusion Criteria:

* Individuals unable to provide 24-hour urine samples.
* Individuals unable to free up a morning for day hospital appointments
* Individuals deprived of liberty by a judicial or administrative decision.
* Adults under a legal protection measure (guardianship, trusteeship).
* Individuals placed under judicial protection.
* Participants enrolled in another study with an ongoing exclusion period
* Pregnant women.
* Individuals not covered by social security

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Urinary oxalate and glycolate excretion | At Day 0
  Comparison of urinary oxalate and glycolate excretion expressed in mmol/L and mmol/24h of symptomatic versus asymptomatic heterozygous AGXT subjects.

SECONDARY OUTCOMES:
The prevalence of stones | At Day 0
  Evaluating the prevalence of stones in asymptomatic heterozygous patients for the AGXT gene using renal ultrasound and through questioning the family history of renal colic or lithiasis and fracture.
Lithiasis disease severity | At Day 0
  Assessing the severity of lithiasis by questioning the frequency of stones and need for urological intervention.
Lithiasis disease severity | At Day 0
  Assessing the severity of lithiasis by using renal ultrasound (size and number of visualized stones)
Lithiasis disease severity | At Day 0
  Assessing the severity of lithiasis by renal function using creatinine level and estimation of glomerular filtration rate (GFR) and Chronic Kidney Disease Epidemiology (CKD-EPI )
Lithiasis disease severity | At Day 0
  Assessing the severity of lithiasis by the number and type of crystals.
Predisposing conditions for lithiasis disease | At Day 0
  Assessing the role of dietary habits in lithiasis disease by using food diary and particularly Fardelonne questionaire.
Predisposing conditions for lithiasis disease | At Day 0
  Assessing the presence of other gene mutations in lithiasis disease using exome sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- CLIMA, pavillon R, Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No